CLINICAL TRIAL: NCT00090753
Title: An Open-label, Multi-center Study to Document the Efficacy, Safety, and Tolerability of Long-term Administration of RO0503821 in Patients With Chronic Renal Anemia
Brief Title: A Study of Intravenous or Subcutaneous Methoxy Polyethylene Glycol-Epoetin Beta (RO0503821, Mircera) in Chronic Kidney Disease Patients With Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH18387
Record Dates: First submitted 2004-09-03; First posted 2004-09-06 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Epoetin Alfa; epoetin beta; Darbepoetin alfa

ARMS (2):
- Methoxy Polyethylene Glycol-Epoetin Beta (Experimental): Patients received the same weekly dose of methoxy polyethylene glycol-epoetin beta via the same route of administration (iv or sc) as they received in the Phase II or Phase III study that qualified the patient for participation in this study. Methoxy polyethylene glycol-epoetin beta was administered every 2 or every 4 weeks in the initial 104-week treatment period. Patients on a 4-week dosing interval were switched to once-monthly administration in the 24-month extension phase. The dose of methoxy polyethylene glycol-epoetin beta was adjusted to maintain the patient's hemoglobin (Hb) within a target range of 11 to 13 g/dL.
  Interventions: Drug: Methoxy Polyethylene Glycol-Epoetin Beta
- Comparator ESA (Active Comparator): Patients received the same comparator ESA [epoetin alfa, epoetin beta, or darbepoetin alfa] at the same weekly dose and dosing interval via the same route of administration (iv or sc) as they received in the Phase III study that qualified the patient for participation in this study. The dose of the comparator drug was adjusted to maintain the patient's Hb within a target range of 11 to 13 g/dL. Of the 480 patients in the comparator drug group, 170 received darbepoetin alfa, 134 received epoetin alfa, and 176 received epoetin beta.
  Interventions: Drug: Epoetin alfa; Drug: Epoetin beta; Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-Epoetin Beta — Methoxy polyethylene glycol-epoetin beta was provided as a sterile single-use injectable solution in 2-mL glass vials containing 1 mL solution or in single-use sterile pre-filled syringes (PFSs) containing 0.3 mL or 0.6 mL injectable solution. The injectable solution was available in vials with the following strengths: 50, 100, 200, 400, and 1000 μg/mL. The injectable solution was available in PFSs with the following strengths: 30, 40, 50, 60, 75, 100, 120, 150, 200, and 250 μg/0.3 mL; and 360 and 400 μg/0.6 mL.
  Other Names: RO0503821; Mircera
  Arms: Methoxy Polyethylene Glycol-Epoetin Beta
Drug: Epoetin alfa — Epoetin alfa was provided with commercial packaging in English with country-specific labels (10,000 IU, 20,000 IU).
  Arms: Comparator ESA
Drug: Epoetin beta — Epoetin beta was provided with commercial packaging in English with country-specific labels (50,000 IU, 100,000 IU).
  Arms: Comparator ESA
Drug: Darbepoetin alfa — Darbepoetin alfa was provided with commercial packaging in English with country-specific labels (vials and PFSs in various strengths).
  Arms: Comparator ESA

SUMMARY:
This study assessed the long-term efficacy, safety, and tolerability of intravenous (iv) or subcutaneous (sc) methoxy polyethylene glycol-epoetin beta in chronic kidney disease patients with renal anemia. Eligible patients were those who were receiving stable maintenance therapy with methoxy polyethylene glycol-epoetin beta or erythropoiesis stimulating agents (ESAs) in Phase II or III clinical studies. They continued to receive methoxy polyethylene glycol-epoetin beta or comparator ESAs at the same weekly dose and by the same route of administration (sc or iv) as in the qualifying studies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult patients (≥ 18 years old) with chronic renal anemia
* Maintenance erythropoietic therapy with methoxy polyethylene glycol-epoetin beta or a protocol-specified reference medication (epoetin alfa formulated with human albumin, epoetin beta or darbepoetin alfa) in one of the following studies: BA16528[NCT00048048], BA16285[NCT00048035], BA16286[NCT00364832], BA16736[NCT00077597], BA16738[NCT00081471], BA16739[NCT00077610], BA16740[NCT00077623], BA17283[NCT00077766] and BA17284[NCT00081484]
* Hemoglobin (Hb) concentration between 10.5 and 13.0 g/dL
* Adequate iron status defined as serum ferritin ≥ 100 ng/mL or Transferrin Saturation (TSAT)≥ 20% or percentage of hypochromic red blood cells (RBCs) < 10%

Exclusion Criteria:

* Poorly controlled hypertension
* History of epileptic seizure
* Pure red cell aplasia
* Chronic congestive heart failure [New York Heart Association (NYHA) IV]
* High likelihood of early withdrawal or interruption of the study
* Active malignant disease (except non-melanoma skin cancer)
* Life expectancy less than 12 months
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2004-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (219):
- United States (72):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Hot Springs, Arkansas
  - Covina, California
  - Encino, California
  - Irvine, California
  - Los Alamitos, California
  - Los Angeles, California
  - Monterey Park, California
  - Mountain View, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Stamford, Connecticut
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Maywood, Illinois
  - South Holland, Illinois
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Brooklyn Center, Minnesota
  - Columbus, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Paterson, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Flushing, New York
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - Orchard Park, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Mount Airy, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Oregon City, Oregon
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Erie, Pennsylvania
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Burlington, Vermont
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Salem, Virginia
  - Morgantown, West Virginia
- Australia (7):
  - Clayton
  - Gosford
  - Liverpool
  - Parkville
  - Perth
  - Sydney
  - Woolloongabba
- Graz, Austria
- Belgium (7):
  - Aalst
  - Brussels
  - Edegem
  - Ghent
  - Hasselt
  - Leuven
  - Liège
- Czechia (3):
  - Liberec
  - Ostrava
  - Pilsen
- Denmark (3):
  - Aalborg
  - Odense
  - Roskilde
- Finland (2):
  - HUS
  - Tampere
- France (25):
  - Bayonne
  - Bois-Guillaume
  - Bordeaux
  - Boulogne
  - Cabestany
  - Caen
  - Chambéry
  - Colmar
  - Hyères
  - La Tronche
  - Limoges
  - Lyon
  - Montpellier
  - Nantes
  - Nîmes
  - Paris
  - Perpignan
  - Poitiers
  - Saint-Germain-en-Laye
  - Saint-Ouen
  - Salouël
  - Tarbes
  - Thionville
  - Toulouse
  - Tours
- Germany (11):
  - Bad Hersfeld
  - Berlin
  - Dortmund
  - Erlangen
  - München
  - Nuremberg
  - Stuttgart
  - Villingen-Schwenningen
  - Wiesbaden
  - Wiesloch
  - Wuppertal
- Greece (5):
  - Alexandroupoli
  - Ioannina
  - Larissa
  - Piraeus
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Debrecen
  - Miskolc
  - Pécs
- Italy (16):
  - Bergamo
  - Cagliari
  - Cremona
  - Cuneo
  - Genova
  - Lecco
  - Livorno
  - Lodi
  - Messina
  - Mestre
  - Modena
  - Pavia
  - Prato
  - Reggio Calabria
  - S Fermo Della Battaglia
  - Venezia
- Mexico (2):
  - Cuernavaca
  - Mexico City
- Heerlen, Netherlands
- Trondheim, Norway
- Panama City, Panama
- Poland (11):
  - Gdansk
  - Gdynia
  - Kielce
  - Krakow
  - Lodz
  - Poznan
  - Rzeszów
  - Szczecin
  - Warsaw
  - Wołomin
  - Wroclaw
- Setúbal, Portugal
- Ponce, Puerto Rico
- Russia (2):
  - Moscow
  - Saint Petersburg
- South Africa (3):
  - Cape Town
  - Durban
  - Soweto
- Spain (18):
  - A Coruña
  - Alcorcón
  - Alicante
  - Almería
  - Badalona
  - Barcelona
  - Bilbao
  - Córdoba
  - L'Hospitalet de Llobregat
  - Lleida
  - Madrid
  - Málaga
  - Oviedo
  - Palma de Mallorca
  - Salamanca
  - Santander
  - Santiago de Compostela
  - Seville
- Sweden (4):
  - Huddinge
  - Karlstad
  - Stockholm
  - Umeå
- Switzerland (2):
  - Aarau
  - Lausanne
- Taiwan (2):
  - Taichung
  - Taipei
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Chon Buri
  - Phitsanulok
- United Kingdom (10):
  - Belfast
  - Cambridge
  - Carshalton
  - Dundee
  - Exeter
  - Glasgow
  - Leicester
  - London
  - Salford
  - Swansea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in one of the following Phase II or Phase III studies: BA16528[NCT00048048], BA16285[NCT00048035], BA16286[NCT00364832], BA16736[NCT00077597], BA16738[NCT00081471], BA16739[NCT00077610], BA16740[NCT00077623], BA17283[NCT00077766] or BA17284[NCT00081484]
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Patients received the same weekly dose of methoxy polyethylene glycol-epoetin beta (Mircera) via the same route of administration (iv or sc) as they received in the Phase II or Phase III study that qualified the patient for participation in this study. Methoxy polyethylene glycol-epoetin beta was administered every 2 or every 4 weeks in the initial 104-week treatment period. Patients on a 4-week dosing interval were switched to once-monthly administration in the 24-month extension phase. The dose of methoxy polyethylene glycol-epoetin beta was adjusted to maintain the patient's hemoglobin (Hb) within a target range of 11 to 13 g/dL.
- Comparator ESA: Patients received the same comparator erythropoiesis stimulating agent (ESA) [epoetin alfa, epoetin beta, or darbepoetin alfa] at the same weekly dose and dosing interval via the same route of administration (iv or sc) as they received in the Phase III study that qualified the patient for participation in this study. The dose of the comparator drug was adjusted to maintain the patient's Hb within a target range of 11 to 13 g/dL. Of the 480 patients in the comparator drug group, 170 received darbepoetin alfa, 134 received epoetin alfa, and 176 received epoetin beta.
Period: First Treatment Period
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta | Comparator ESA
Started | 748 | 480
Completed | 492 | 302
Not Completed | 256 | 178
Not completed — Adverse Event | 20 | 8
Not completed — Death | 88 | 62
Not completed — Lack of Efficacy | 2 | 1
Not completed — Refused Treatment | 32 | 25
Not completed — Lost to Follow-up | 4 | 4
Not completed — Renal Transplant | 70 | 50
Not completed — Mircera Commercialization | 1 | 0
Not completed — Other Unrelated to Safety and Efficacy | 39 | 28
Period: Extended Treatment Period
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta | Comparator ESA
Started | 453 (39 patients who completed the first treatment period refused to enter the extended treatment period.) | 250 (52 patients who completed the first treatment period refused to enter the extended treatment period.)
Completed | 94 | 59
Not Completed | 359 | 191
Not completed — Adverse Event | 11 | 0
Not completed — Death | 58 | 30
Not completed — Lack of Efficacy | 1 | 0
Not completed — Refused Treatment | 18 | 12
Not completed — Lost to Follow-up | 3 | 1
Not completed — Renal Transplant | 15 | 12
Not completed — Mircera Commercialization | 188 | 93
Not completed — Other Unrelated to Safety and Efficacy | 65 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta | Comparator ESA | Total
Number analyzed (Participants) | 748 | 480 | 1228
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (14.80) | 61.9 (14.42) | 61.5 (14.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 223 | 550
  Male | 421 | 257 | 678

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin Concentration to the Last Month of Study Participation
Description: Blood samples were collected at each study visit, that is, every 4 weeks for the first 12 weeks, every 12 weeks until week 105 of the first study period, every 3 months thereafter, and at the end of study or the last visit if the patient discontinued the study prematurely.
Time Frame: Baseline to the end of the study (Up to 49 Months)
Population: Analysis includes participants from the Intent-to-treat population (all patients who received at least 1 dose of methoxy polyethylene glycol-epoetin beta or a comparator ESA) who had hemoglobin values available for analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta | Comparator ESA
Number analyzed (Participants) | 735 | 476
g/dL | -0.55 (1.832) | -0.38 (1.614)

2. Secondary Outcome: Percentage of Patients Who Had at Least 1 Adverse Event
Description: See the adverse events section of the results for more information.
Time Frame: From first dose of study drug to date of last contact or 30 days after last drug dose (Up to 49 months)
Population: Intent-to-treat population: All patients who received at least 1 dose of methoxy polyethylene glycol-epoetin beta or a comparator ESA.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta | Comparator ESA
Number analyzed (Participants) | 748 | 480
Percentage of participants | 94.3 | 93.3

ADVERSE EVENTS:
Time Frame: From first dose of study drug to date of last contact or 30 days after last drug dose (Up to 49 months)
Description: Intent-to-treat population: All patients who received at least 1 dose of methoxy polyethylene glycol-epoetin beta or a comparator ESA.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta | Comparator ESA
Serious Adverse Events (participants affected / at risk) | 499/748 | 316/480
Other Adverse Events (participants affected / at risk) | 624/748 | 390/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=748) | Comparator ESA (N=480)
PNEUMONIA (Infections and infestations) | 53 | 35
SEPSIS (Infections and infestations) | 24 | 12
CELLULITIS (Infections and infestations) | 15 | 7
BRONCHITIS (Infections and infestations) | 10 | 8
GASTROENTERITIS (Infections and infestations) | 11 | 4
CATHETER SEPSIS (Infections and infestations) | 7 | 6
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 7 | 5
GANGRENE (Infections and infestations) | 7 | 5
SEPTIC SHOCK (Infections and infestations) | 8 | 4
BRONCHOPNEUMONIA (Infections and infestations) | 6 | 5
CATHETER RELATED INFECTION (Infections and infestations) | 8 | 3
URINARY TRACT INFECTION (Infections and infestations) | 7 | 4
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 6 | 4
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 5 | 4
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 6 | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 5 | 3
OSTEOMYELITIS (Infections and infestations) | 5 | 3
DIABETIC GANGRENE (Infections and infestations) | 5 | 2
DIVERTICULITIS (Infections and infestations) | 6 | 1
CENTRAL LINE INFECTION (Infections and infestations) | 4 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 2
APPENDICITIS (Infections and infestations) | 4 | 1
ARTERIOVENOUS FISTULA SITE INFECTION (Infections and infestations) | 1 | 4
ENDOCARDITIS (Infections and infestations) | 3 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 3 | 2
UROSEPSIS (Infections and infestations) | 4 | 1
INFECTED SKIN ULCER (Infections and infestations) | 4 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 3
WOUND INFECTION (Infections and infestations) | 3 | 1
BACTERAEMIA (Infections and infestations) | 2 | 1
CATHETER BACTERAEMIA (Infections and infestations) | 3 | 0
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 2 | 1
DIABETIC FOOT INFECTION (Infections and infestations) | 1 | 2
INTERVERTEBRAL DISCITIS (Infections and infestations) | 2 | 1
LUNG INFECTION (Infections and infestations) | 2 | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 1
BACTERIAL INFECTION (Infections and infestations) | 2 | 0
BACTERIAL SEPSIS (Infections and infestations) | 1 | 1
CATHETER SITE INFECTION (Infections and infestations) | 2 | 0
CELLULITIS GANGRENOUS (Infections and infestations) | 2 | 0
ERYSIPELAS (Infections and infestations) | 0 | 2
FUNGAEMIA (Infections and infestations) | 2 | 0
GRAFT INFECTION (Infections and infestations) | 1 | 1
GROIN ABSCESS (Infections and infestations) | 1 | 1
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 2 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 2 | 0
PYELONEPHRITIS (Infections and infestations) | 2 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 1
ABDOMINAL SEPSIS (Infections and infestations) | 0 | 1
ANOGENITAL WARTS (Infections and infestations) | 1 | 0
ARTERIOSCLEROTIC GANGRENE (Infections and infestations) | 0 | 1
ARTERITIS INFECTIVE (Infections and infestations) | 0 | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 1
BACTERIAL DIARRHOEA (Infections and infestations) | 0 | 1
BALANOPOSTHITIS INFECTIVE (Infections and infestations) | 1 | 0
CELLULITIS OF MALE EXTERNAL (Infections and infestations) | 1 | 0
GENITAL ORGAN CELLULITIS STREPTOCOCCAL (Infections and infestations) | 1 | 0
CHRONIC TONSILLITIS (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 | 1
EMPHYSEMATOUS CHOLECYSTITIS (Infections and infestations) | 1 | 0
EMPYEMA (Infections and infestations) | 1 | 0
ENDOCARDITIS STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
EYE INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
FUNGAL PERITONITIS (Infections and infestations) | 0 | 1
GASTRIC ULCER HELICOBACTER (Infections and infestations) | 0 | 1
HAEMATOMA INFECTION (Infections and infestations) | 0 | 1
HEPATITIS C (Infections and infestations) | 1 | 0
INFECTED BITES (Infections and infestations) | 1 | 0
INFECTED CYST (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0
KLEBSIELLA SEPSIS (Infections and infestations) | 1 | 0
LIVER ABSCESS (Infections and infestations) | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
NOSOCOMIAL INFECTION (Infections and infestations) | 1 | 0
ORAL INFECTION (Infections and infestations) | 0 | 1
OSTEOMYELITIS CHRONIC (Infections and infestations) | 0 | 1
PANCREAS INFECTION (Infections and infestations) | 0 | 1
PAROTID ABSCESS (Infections and infestations) | 1 | 0
PHARYNGEAL ABSCESS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 0
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 | 0
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1
POST PROCEDURAL SEPSIS (Infections and infestations) | 1 | 0
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 1 | 0
PULMONARY SEPSIS (Infections and infestations) | 0 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 | 0
RECTAL ABSCESS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 1
SEPTIC ARTHRITIS STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
SERRATIA BACTERAEMIA (Infections and infestations) | 1 | 0
SERRATIA INFECTION (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL OSTEOMYELITIS (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1
TUBERCULOSIS (Infections and infestations) | 1 | 0
TUBERCULOUS PLEURISY (Infections and infestations) | 1 | 0
WEST NILE VIRAL INFECTION (Infections and infestations) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 27 | 15
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 19 | 21
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 26 | 10
ATRIAL FIBRILLATION (Cardiac disorders) | 16 | 19
CARDIAC ARREST (Cardiac disorders) | 16 | 11
ANGINA PECTORIS (Cardiac disorders) | 16 | 9
CORONARY ARTERY DISEASE (Cardiac disorders) | 9 | 9
ACUTE CORONARY SYNDROME (Cardiac disorders) | 10 | 3
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 5 | 6
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 7 | 4
ATRIAL FLUTTER (Cardiac disorders) | 7 | 3
VENTRICULAR FIBRILLATION (Cardiac disorders) | 6 | 4
BRADYCARDIA (Cardiac disorders) | 8 | 1
CARDIAC FAILURE (Cardiac disorders) | 5 | 3
ARRHYTHMIA (Cardiac disorders) | 4 | 2
CARDIOGENIC SHOCK (Cardiac disorders) | 4 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 4 | 1
ANGINA UNSTABLE (Cardiac disorders) | 4 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 3
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 3
PERICARDITIS (Cardiac disorders) | 3 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 3 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 2 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 1
TACHYCARDIA (Cardiac disorders) | 2 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 | 1
COR PULMONALE (Cardiac disorders) | 2 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 1
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 2 | 0
PALPITATIONS (Cardiac disorders) | 1 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 1 | 1
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR DISSOCIATION (Cardiac disorders) | 1 | 0
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISSECTION (Cardiac disorders) | 1 | 0
ELECTROMECHANICAL DISSOCIATION (Cardiac disorders) | 0 | 1
HYPERTENSIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 | 0
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1 | 0
NODAL ARRHYTHMIA (Cardiac disorders) | 1 | 0
PERICARDIAL DISEASE (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
SINUS ARRHYTHMIA (Cardiac disorders) | 1 | 0
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1 | 0
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 26 | 20
ARTERIOVENOUS GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 16 | 8
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 6 | 9
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 11 | 3
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 7 | 4
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 9 | 2
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 6 | 4
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 5 | 4
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 7 | 2
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 3 | 6
HIP FRACTURE (Injury, poisoning and procedural complications) | 5 | 3
ARTERIOVENOUS FISTULA ANEURYSM (Injury, poisoning and procedural complications) | 4 | 3
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 5 | 2
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 2 | 3
ARTERIOVENOUS GRAFT SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 3 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 2 | 2
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 | 2
HEAD INJURY (Injury, poisoning and procedural complications) | 2 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 2 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 2 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
CONCUSSION (Injury, poisoning and procedural complications) | 2 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 2
JOINT INJURY (Injury, poisoning and procedural complications) | 2 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 2 | 0
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 2
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 0 | 2
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
ARTERIOVENOUS FISTULA OCCLUSION (Injury, poisoning and procedural complications) | 0 | 1
ARTERIOVENOUS FISTULA SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
ARTERIOVENOUS GRAFT ANEURYSM (Injury, poisoning and procedural complications) | 0 | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 1 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
DELAYED RECOVERY FROM ANAESTHESIA (Injury, poisoning and procedural complications) | 0 | 1
DEVICE MALFUNCTION (Injury, poisoning and procedural complications) | 0 | 1
DIALYSIS DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FRACTURED COCCYX (Injury, poisoning and procedural complications) | 0 | 1
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
PERIRENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL PULMONARY EMBOLISM (Injury, poisoning and procedural complications) | 0 | 1
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 0 | 1
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1 | 0
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 | 1
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UROSTOMY COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 8 | 8
PERITONITIS (Gastrointestinal disorders) | 8 | 6
GASTRITIS (Gastrointestinal disorders) | 9 | 3
DIARRHOEA (Gastrointestinal disorders) | 7 | 4
PANCREATITIS (Gastrointestinal disorders) | 8 | 2
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 5 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 4
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 4 | 2
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 4 | 2
VOMITING (Gastrointestinal disorders) | 4 | 2
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 5 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 2
COLITIS (Gastrointestinal disorders) | 3 | 1
COLONIC POLYP (Gastrointestinal disorders) | 3 | 1
INTESTINAL INFARCTION (Gastrointestinal disorders) | 2 | 2
MELAENA (Gastrointestinal disorders) | 2 | 2
ABDOMINAL HERNIA (Gastrointestinal disorders) | 2 | 1
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 | 2
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
DUODENITIS (Gastrointestinal disorders) | 3 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 3
ILEUS (Gastrointestinal disorders) | 2 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 2
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 2 | 0
CAECITIS (Gastrointestinal disorders) | 0 | 2
DIVERTICULUM (Gastrointestinal disorders) | 0 | 2
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 2 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 1
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 2 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 1 | 1
REFLUX OESOPHAGITIS (Gastrointestinal disorders) | 2 | 0
SUBILEUS (Gastrointestinal disorders) | 1 | 1
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
DIVERTICULITIS INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 1 | 0
DUODENITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
EROSIVE DUODENITIS (Gastrointestinal disorders) | 0 | 1
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 1
GASTRIC DISORDER (Gastrointestinal disorders) | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0
GASTRODUODENITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL TELANGIECTASIA (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
MEGACOLON (Gastrointestinal disorders) | 1 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0
RETROPERITONEAL FIBROSIS (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 7 | 8
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 6 | 6
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 8 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 5 | 3
CEREBRAL INFARCTION (Nervous system disorders) | 4 | 3
SYNCOPE (Nervous system disorders) | 5 | 2
CAROTID ARTERY STENOSIS (Nervous system disorders) | 5 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 5 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 4 | 1
CEREBROVASCULAR DISORDER (Nervous system disorders) | 3 | 1
CONVULSION (Nervous system disorders) | 3 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 3 | 0
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 2 | 1
PRESYNCOPE (Nervous system disorders) | 2 | 1
DIZZINESS (Nervous system disorders) | 2 | 0
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 1
EMBOLIC STROKE (Nervous system disorders) | 1 | 1
EPILEPSY (Nervous system disorders) | 0 | 2
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 1 | 1
HYPOGLYCAEMIC COMA (Nervous system disorders) | 2 | 0
HYPOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 1
LACUNAR INFARCTION (Nervous system disorders) | 1 | 1
REVERSIBLE ISCHAEMIC NEUROLOGICAL DEFICIT (Nervous system disorders) | 1 | 1
URAEMIC NEUROPATHY (Nervous system disorders) | 2 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
ANOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
BALANCE DISORDER (Nervous system disorders) | 1 | 0
BENIGN INTRACRANIAL HYPERTENSION (Nervous system disorders) | 1 | 0
CEREBRAL ARTERIOSCLEROSIS (Nervous system disorders) | 0 | 1
CEREBRAL ATROPHY (Nervous system disorders) | 1 | 0
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0
COMA HEPATIC (Nervous system disorders) | 1 | 0
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 1 | 0
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 | 0
DEMENTIA WITH LEWY BODIES (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
HAEMORRHAGIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 0 | 1
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
MUSCLE SPASTICITY (Nervous system disorders) | 0 | 1
NEURALGIA (Nervous system disorders) | 1 | 0
NEUROTOXICITY (Nervous system disorders) | 0 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 1 | 0
POLYNEUROPATHY (Nervous system disorders) | 1 | 0
SENILE DEMENTIA (Nervous system disorders) | 0 | 1
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 1 | 0
STUPOR (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 12 | 6
HYPERTENSION (Vascular disorders) | 9 | 6
PERIPHERAL ISCHAEMIA (Vascular disorders) | 7 | 6
DEEP VEIN THROMBOSIS (Vascular disorders) | 5 | 2
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 4 | 3
DIABETIC VASCULAR DISORDER (Vascular disorders) | 4 | 2
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 4 | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 2 | 3
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 4 | 0
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 3 | 1
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 3 | 0
ARTERIAL STENOSIS LIMB (Vascular disorders) | 1 | 2
HYPERTENSIVE EMERGENCY (Vascular disorders) | 2 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 | 1
VENOUS STENOSIS (Vascular disorders) | 1 | 2
ACCELERATED HYPERTENSION (Vascular disorders) | 2 | 0
AORTIC STENOSIS (Vascular disorders) | 1 | 1
ARTERIAL STENOSIS (Vascular disorders) | 0 | 2
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 1
ARTERIOSCLEROSIS OBLITERANS (Vascular disorders) | 2 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 2 | 0
EXTREMITY NECROSIS (Vascular disorders) | 2 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 2 | 0
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 2
STEAL SYNDROME (Vascular disorders) | 1 | 1
ANEURYSM (Vascular disorders) | 0 | 1
ANEURYSM RUPTURED (Vascular disorders) | 0 | 1
ANGIOPATHY (Vascular disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 1 | 0
AORTIC DISSECTION (Vascular disorders) | 0 | 1
ARTERIAL DISORDER (Vascular disorders) | 1 | 0
BRACHIOCEPHALIC VEIN STENOSIS (Vascular disorders) | 1 | 0
FEMORAL ARTERY EMBOLISM (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 1
ISCHAEMIA (Vascular disorders) | 0 | 1
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 1
MICROANGIOPATHY (Vascular disorders) | 0 | 1
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 | 0
PHLEBITIS (Vascular disorders) | 1 | 0
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 | 0
VASCULAR CALCIFICATION (Vascular disorders) | 1 | 0
VASCULAR RUPTURE (Vascular disorders) | 1 | 0
VASCULAR STENOSIS (Vascular disorders) | 0 | 1
VASCULITIS (Vascular disorders) | 1 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 1 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 9 | 12
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 10 | 7
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 6 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 3
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 6 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 5 | 2
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 | 3
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 0
NON-CARDIOGENIC PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
MEDIASTINAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY VASCULITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
TRACHEAL ULCER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
WEGENER'S GRANULOMATOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 16 | 11
HYPERKALAEMIA (Metabolism and nutrition disorders) | 15 | 12
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 7 | 10
DIABETIC FOOT (Metabolism and nutrition disorders) | 3 | 7
CACHEXIA (Metabolism and nutrition disorders) | 4 | 5
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 4 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 2
GOUT (Metabolism and nutrition disorders) | 3 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 | 1
CALCIPHYLAXIS (Metabolism and nutrition disorders) | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 1
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
DEATH (General disorders) | 7 | 8
PYREXIA (General disorders) | 10 | 5
NON-CARDIAC CHEST PAIN (General disorders) | 9 | 4
CATHETER THROMBOSIS (General disorders) | 3 | 4
SUDDEN DEATH (General disorders) | 2 | 4
CATHETER RELATED COMPLICATION (General disorders) | 2 | 3
CHEST PAIN (General disorders) | 2 | 2
MULTI-ORGAN FAILURE (General disorders) | 2 | 2
ASTHENIA (General disorders) | 2 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 | 0
HYPERPYREXIA (General disorders) | 3 | 0
HERNIA OBSTRUCTIVE (General disorders) | 2 | 0
HYPERTHERMIA (General disorders) | 1 | 1
SUDDEN CARDIAC DEATH (General disorders) | 2 | 0
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 2 | 0
CALCINOSIS (General disorders) | 1 | 0
CATHETER SITE HAEMORRHAGE (General disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0
CHILLS (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 0 | 1
IMPLANT SITE NECROSIS (General disorders) | 0 | 1
INFLAMMATION (General disorders) | 0 | 1
MULTI-ORGAN DISORDER (General disorders) | 0 | 1
OEDEMA DUE TO RENAL DISEASE (General disorders) | 0 | 1
PAIN (General disorders) | 1 | 0
PSEUDOCYST (General disorders) | 0 | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 22 | 15
RENAL FAILURE ACUTE (Renal and urinary disorders) | 4 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 3
AZOTAEMIA (Renal and urinary disorders) | 2 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 2
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 0
NEPHROPATHY TOXIC (Renal and urinary disorders) | 1 | 0
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 1 | 0
PYELOCALIECTASIS (Renal and urinary disorders) | 0 | 1
RENAL CYST RUPTURED (Renal and urinary disorders) | 1 | 0
RENAL DISORDER (Renal and urinary disorders) | 0 | 1
RENAL HAEMORRHAGE (Renal and urinary disorders) | 1 | 0
RENAL HYPERTENSION (Renal and urinary disorders) | 0 | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 | 1
URINARY BLADDER POLYP (Renal and urinary disorders) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
ADENOID CYSTIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PARATHYROID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
URINARY TRACT NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
DACTYLITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEODYSTROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 15 | 6
HYPERPARATHYROIDISM TERTIARY (Endocrine disorders) | 2 | 2
HYPERPARATHYROIDISM (Endocrine disorders) | 1 | 2
HYPERTHYROIDISM (Endocrine disorders) | 1 | 1
GOITRE (Endocrine disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 7 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 4 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 3 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0
GALLBLADDER POLYP (Hepatobiliary disorders) | 1 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0
HEPATIC CONGESTION (Hepatobiliary disorders) | 1 | 0
HEPATIC FIBROSIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 1 | 0
HEPATOSPLENOMEGALY (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 4 | 5
CONFUSIONAL STATE (Psychiatric disorders) | 3 | 1
ANXIETY (Psychiatric disorders) | 2 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 | 0
ANXIETY DISORDER (Psychiatric disorders) | 1 | 0
BIPOLAR I DISORDER (Psychiatric disorders) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
DELIRIUM (Psychiatric disorders) | 0 | 1
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 | 1
DISORIENTATION (Psychiatric disorders) | 0 | 1
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 9 | 3
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 3 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2 | 0
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 2 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETIC NEUROPATHIC ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 0 | 1
PENILE ULCERATION (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 10 | 6
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
HYPOPROTHROMBINAEMIA (Blood and lymphatic system disorders) | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
CATARACT (Eye disorders) | 3 | 4
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 | 0
GLAUCOMA (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
CERVIX INFLAMMATION (Reproductive system and breast disorders) | 0 | 1
CYSTOCELE (Reproductive system and breast disorders) | 1 | 0
GENITAL PROLAPSE (Reproductive system and breast disorders) | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1
PROSTATISM (Reproductive system and breast disorders) | 1 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
TESTICULAR INFARCTION (Reproductive system and breast disorders) | 0 | 1
UTERINE CERVICAL SQUAMOUS METAPLASIA (Reproductive system and breast disorders) | 0 | 1
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 0 | 3
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
ANAPHYLACTOID REACTION (Immune system disorders) | 0 | 1
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Congenital, familial and genetic disorders) | 2 | 0
CONGENITAL CYSTIC KIDNEY DISEASE (Congenital, familial and genetic disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 2
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 1
BACTERIAL CULTURE POSITIVE (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=748) | Comparator ESA (N=480)
NASOPHARYNGITIS (Infections and infestations) | 107 | 64
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 81 | 63
URINARY TRACT INFECTION (Infections and infestations) | 77 | 57
BRONCHITIS (Infections and infestations) | 75 | 49
INFLUENZA (Infections and infestations) | 48 | 23
GASTROENTERITIS (Infections and infestations) | 33 | 27
DIARRHOEA (Gastrointestinal disorders) | 141 | 96
VOMITING (Gastrointestinal disorders) | 73 | 44
NAUSEA (Gastrointestinal disorders) | 59 | 41
CONSTIPATION (Gastrointestinal disorders) | 52 | 41
ABDOMINAL PAIN (Gastrointestinal disorders) | 46 | 22
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 37 | 27
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 75 | 56
BACK PAIN (Musculoskeletal and connective tissue disorders) | 74 | 44
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 76 | 41
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 65 | 42
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 55 | 30
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 44 | 24
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 97 | 56
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 83 | 36
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 56 | 24
ARTERIOVENOUS GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 53 | 26
CONTUSION (Injury, poisoning and procedural complications) | 34 | 27
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 39 | 22
HYPERTENSION (Vascular disorders) | 167 | 109
HYPOTENSION (Vascular disorders) | 31 | 26
FLUID OVERLOAD (Metabolism and nutrition disorders) | 83 | 38
HYPERKALAEMIA (Metabolism and nutrition disorders) | 47 | 37
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 47 | 22
COUGH (Respiratory, thoracic and mediastinal disorders) | 79 | 58
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 62 | 41
HEADACHE (Nervous system disorders) | 83 | 43
INSOMNIA (Psychiatric disorders) | 39 | 33
DEPRESSION (Psychiatric disorders) | 38 | 21
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 57 | 44
PRURITUS (Skin and subcutaneous tissue disorders) | 59 | 35
PYREXIA (General disorders) | 52 | 27
ATRIAL FIBRILLATION (Cardiac disorders) | 42 | 30
ANAEMIA (Blood and lymphatic system disorders) | 41 | 25
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 22 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights